CLINICAL TRIAL: NCT00831467
Title: Safety and Efficacy Trial of a RNActive®-Derived Prostate Cancer Vaccine in Hormone Refractory Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CureVac (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CV-9103-001
Record Dates: First submitted 2009-01-27; First posted 2009-01-29 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Hormonal Refractory Prostate Cancer
Keywords: Hormonal refractory prostate cancer; RNA vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CV9103 (Experimental): CV9103 is applied intradermally into the thigh and upper arm of either side of the body at week 1, week 3, week 7, week 15, week 23
  Interventions: Biological: CV9103

INTERVENTIONS:
Biological: CV9103 — Over a period of 23 weeks 5 vaccinations with CV9103 will be administered.

SUMMARY:
The purpose of this study is to determine the efficacy and safety of a new vaccine in hormone refractory prostate cancer

DETAILED DESCRIPTION:
Immunotherapy of prostate cancer is a promising approach for the treatment of advanced or recurrent forms of prostate cancer. Recently, immunotherapy of prostate cancer has been facilitated by the identification of a number of prostate specific antigens that are expressed in healthy and tumor prostate tissues. For prostatectomized patients, such antigens offer ideal targets for immunotherapy as they are only present in tumor but not in healthy tissue. The use of prostate specific antigens in a cancer vaccine is one attractive option for cancer immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent in accordance with GCP and local regulatory requirements prior to trial participation
* Male and age ≥ 18 years (Phase I and II) and ≤ 75 years (Phase II only)
* Histologically confirmed diagnosis of adenocarcinoma of the prostate, Gleason Score available
* Patients must have been treated with hormonal therapy and may have been treated with surgery and/ or radiation therapy
* Progressive disease as defined by hormone-refractoriness and rise in PSA:

Hormone-refractoriness: Defined by a rise in PSA and/or RECIST-based progression of evaluable lesions, and/or increased number of hotspots on a bone scan, while the patient has a castrated level of testosterone. This castrated level may have been obtained by orchiectomy, or LH-RH analog ± antiandrogen. Antiandrogen must be discontinued for at least 4 weeks before study entry to exclude a withdrawal effect.

Rise in PSA: Defined by a rise in PSA levels at three consecutive time points (PSA rise over nadir, separated by > 1 week, PCWG2 criteria)

* Presence of metastatic disease is acceptable
* ECOG performance status of 0 to 1
* Life expectancy > 12 months as assessed by the investigator
* Adequate organ function :

Bone marrow function: Hemoglobin ≥ 10 g/dL; Leukocytes ≥ 3000/µL; Lymphocytes ≥ 1000/µL; Absolute neutrophil count ≥ 1500/µL; Platelet count ≥ 100000/µL Hepatic: AST and ALT ≤ 2.5 times upper limit of normal (ULN); Bilirubin ≤ 1.5 ULN Renal: Creatinine ≤ 1.5 mg/dL or creatinine clearance ≥ 60mL/min

* Concomitant LH-RH therapy continuation is acceptable
* May have had local palliative radiotherapy for bone metastasis involving less than 25% of bone marrow
* Patients requiring bisphosphonates at the time of registration into the trial are eligible (therapy initiated at least 28 days prior to first study treatment administration) and must be continued at a constant level during the study period.
* Patients of child-producing potential must agree to use contraception while enrolled in the study and for one month after the last immunization.

Exclusion Criteria:

* Other histologic type of prostate cancer (transitional cell, small cell or squamous cell cancer)
* Symptomatic brain metastasis or leptomeningeal involvement
* Patients having received or currently receiving chemo- or biological therapy for prostate cancer
* Symptomatic congestive heart failure (NYHA 3 and 4); unstable angina pectoris; significant cardiac arrhythmia
* Pulmonary disease causing dyspnea or fatigue during normal activity
* History of seizures, encephalitis or multiple sclerosis
* Inflammatory bowel disease e.g. Crohn's disease or ulcerative colitis; active diverticulitis
* Documented history of active autoimmune disorders requiring systemic immunosuppressive therapy, (e.g. sarcoidosis, lupus erythematosus, rheumatoid arthritis, glomerulonephritis or systemic vasculitis), excepting autoimmune thyroiditis with only thyroid hormone replacement and stable disease > 1 year
* Primary or secondary immune deficiency
* History of allergy requiring medication
* Active drug abuse or chronic alcoholism
* Clinically significant active infections
* Seropositive for HIV, HBV or HCV
* History of other malignancies over the last 5 years (except basal cell carcinoma of the skin)
* Uncontrolled medical condition considered as high risk for the treatment with an investigational drug including unstable diabetes mellitus, vena-cava-syndrome, known ascites and/or pleural effusion, symptomatic pleural effusion treated by puncture
* Renal insufficiency requiring dialysis
* Patients being committed to an institution by virtue of an order issued either by the judicial or the administrative authorities

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2009-01; Primary Completion 2009-12 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Determination of the recommended dose for exploration in the phase II part | 6-9 months
Assessment of Safety of trial regimen | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Miller, Professor, Principal Investigator — PMID: 19143027
Locations (12):
- Germany (11):
  - Universitätsklinikum Aachen, Urologische Klinik, Aachen
  - Charité Universitätsmedizin Berlin, Urologische Klinik u. Hochschulambulanz, Berlin
  - Universitätsklinikum Carl Gustav Carus der TU Dresden, Klinik und Poliklinik für Urologie, Dresden
  - Universitätsklinikum Essen, Klinik und Poliklinik für Urologie, Uroonkologie und Kinderurologie, Essen
  - Klinikum der JWG-Universität, Klinik für Urologie und Kinderurologie, Frankfurt am Main
  - Universitätsklinikum Freiburg, Abteilung Urologie, Freiburg im Breisgau
  - UKSH Campus Lübeck, Klinik und Poliklinik fur Urologie, Lübeck
  - Johannes-Gutenberg-Universität Mainz, Urologische Klinik und Poliklinik, Mainz
  - Universitätsmedizin Mannheim, Urologische Klinik, Mannheim
  - Klinikum rechts der Isar der TU München, Urologische Klinik und Poliklinik, München
  - Klinik für Urologie, Universitätsklinikum Tübingen, Tübingen
- Fondazione scientifica Istituto San Raffaele, Milan, Italy

REFERENCES:
- [Derived] Fotin-Mleczek M, Duchardt KM, Lorenz C, Pfeiffer R, Ojkic-Zrna S, Probst J, Kallen KJ. Messenger RNA-based vaccines with dual activity induce balanced TLR-7 dependent adaptive immune responses and provide antitumor activity. J Immunother. 2011 Jan;34(1):1-15. doi: 10.1097/CJI.0b013e3181f7dbe8. PMID 21150709